CLINICAL TRIAL: NCT05682911
Title: Hypolipidemic, Cardioprotective and Antioxidant Effect of Zingiber Officinale L. Extract in Hypertensive Patients: A Clinical Approach
Brief Title: Protective Effect of Zingiber Officinale L. Extract in Hypertensive Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jinnah Sindh Medical University (Other)
Collaborators: Al Khidmat Hospital Nazimabad Karachi (Unknown); Medics Laboratories (Pvt.) Ltd. (Unknown)
Responsible Party: Principal Investigator, sadaf naeem, Associate Professor, Jinnah Sindh Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 026-HV/HP-2017
Record Dates: First submitted 2022-11-26; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: The Main Focus of This Study is to Evaluate the Safety of Zingiber Officinale L. Tablets as Hypolipidemic Agent in Hypertensive Patients
Keywords: Zingiber officinale L., Hyperlipidemia, Clinical study,Cardioprotective, Antioxidant
MeSH Terms: conditions — Hyperlipidemias | interventions — ginger extract; Simvastatin

STUDY DESIGN:
Intervention Model Description: A two-arm parallel assignment involves two groups of participants. One group receives simvastatin 20mg OD, and the other group receives 500mg Ginger extract tablet BD.
Who Masked: Participant, Care Provider
Masking Description: Blinding was maintained by keeping identical packaging of the ginger and simvastatin drugs with different codes, and no aroma was detected from either; the participants and their care giver were blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zingiber Officinale L (Ginger) treated group n=20 (Experimental): Ginger tablets 500mg twice a day (BD) for two month
  Interventions: Drug: Zingiber officinale L. tablets
- Simvastatin treated group n=20 (Active Comparator): Simvastatin 20 mg tablet once a day (OD) for two month
  Interventions: Drug: Simvastatin 20mg

INTERVENTIONS:
Drug: Zingiber officinale L. tablets — Zingiber officinale L. tablets 500mg twice daily
  Other Names: Ginger tablets
  Arms: Zingiber Officinale L (Ginger) treated group n=20
Drug: Simvastatin 20mg — Simvastatin 20mg once a day for 2 months
  Other Names: Limitrol 20mg
  Arms: Simvastatin treated group n=20

SUMMARY:
Hyperlipidemia is a well-known risk factor for cardiovascular diseases (CVDs). Coronary heart disease, stroke, and atherosclerosis are among the primary cause of death. Various medicines are available for the treatment of hyperlipidemia however, they are linked with serious unwanted effects. Zingiber officinale L. extract (Ginger) was used in folklore medicine as a hypolipidemic agent, Although, its clinical trial studies were not been investigated in the Pakistani population yet. Our clinical study is the first to assess the hypolipidemic, antioxidant, and cardioprotective effect of ginger tablets on dyslipidemic patients regarded as important risk factors for cardiovascular morbidity. A total of 40 dyslipidemic patients of age (18-65 years) of either sex were recruited in Al-Khidmat Hospital Karachi and allocated into two groups; the Simvastatin group (20 mg OD) and the Ginger treated group (500mg Ginger tablets BD) for 2 months. At baseline, their Blood pressure (BP), heart rate (HR), Insomnia severity index (ISI), Minimental state examination (MMSE), Lipid profile, Serum Glutamic Oxaloacetic Transaminase (SGOT), Serum Glutamic Pyruvic Transaminase (SGPT), creatine kinase (CK-MB), C-reactive protein, Superoxide Dismutase (SOD) & Glutathione Peroxidase (GPx) were recorded and repeated after 2 months of follow-up.

DETAILED DESCRIPTION:
1. Study area and setting The study covered the period of January, 2018 to June, 2018 in the Al-Khidmat Medical and Diagnostic Center Nazimabad No.2, Karachi. This was carried out with the cooperation of Cardiac OPD and Laboratory Department of Al-Khidmat Medical and Diagnostic Center. All procedures were approved by the Independent Ethics Committee (IEC) of International Center for Chemical and Biological Sciences (ICCBS), University of Karachi (Study Number. 026-HV/HP-2017, Protocol Number. ICCBS/IEC-026-HV/HP-2017/Protocol/2.0) dated December 08, 2017.
2. Study design This was single blind randomized clinical Study of 40 hyperlipidemic patients. The determination of sample size was done on basis of data from past studies and calculated from formula on SPSS. All the newly diagnosed hyperlipidemic patients were recruited according to the inclusion and exclusion criteria. the written informed consent in local language was being taken to all before the study. The questionnaires used to record information related to the demographic profile, age, gender, family history, past medical history, past laboratory findings, diagnosis and current treatment. All pateints were examined with blood pressure, pulse rate, total lipid profile and cardio-vascular biomarker.
3. Selection of participants A total 40 newly diagnosed hyperlipidemic patients visiting Cardiac OPD at Al-Khidmat Medical and Diagnostic Center, Nazimabad No. 2 Karachi were selected for this study on basis of inclusion and exclusion criteria. Patients were randomized (1:1) using a computer-generated table into two groups: the control group received simvastatin and treated group powder tablets twice a day. Ginger treated group was treated with ginger powder tablets 500mg twice a day (BD) for two month while Simvastatin treated group was maintained on simvastatin 20 mg tablet once a day (OD) for two month. All the patients were over eighteen years of age, conversant in Urdu, consented to be available for participation in eight week study (Two months). The duration of treatment was decided on basis of previous studies carried.

   The inclusion criteria included patients were above 18 years age, either male or female with the diagnosis of hyperlipidemia, total cholesterol up to 200-239mg/dl and LDL 100-159mg/dl. They must not receive lipid-lowering drugs for at least 3 months prior to the recruitment and clinical laboratory tests (CBC, Blood Chemistry, and Urinalysis) were within normal ranges. Exclusions criteria were any cardiovascular diseases, seizures, previous liver surgery, poor controlled diabetes, and drug/alcohol dependence, pregnancy and GI ulcer. Subjects receiving antihyperlipidemic agents (Statins, Niacin, Fibrates and Bile Sequestrants) were excluded in recent past. Blinding was maintained by keeping identical packaging of the ginger and simvastatin drugs with different codes, and no aroma was detected from either; the participants were blinded to the treatment allocation.
4. Study protocol Patients that met the above criteria and gave written consent were randomized to the Treatment group (ginger tablet) and the Control group (Simvastatin) for 8 weeks. During the initial evaluations, all patients interviewed by taking patients previous history included the questions about medical illness, medications, allergies and family history of illness and disease status, blood pressure and pulse rate on every visit. Blood sample (5 ml) was taken before and after treatment for total Lipid Profile, SGPT, SGOT, CK-MB and C-RP. Erythrocyte antioxidant enzymes activity of superoxide dismutase (SOD) and glutathione peroxidase (GPX) were determined by spectrometric method using Ransod and Ransel kit, respectively. Upon every visit all patients were also screened with their blood pressures, heart rate, sleep pattern by insomnia severity indexed (26) and memory by MMSE (27). Analysis was blinded and was performed at the same laboratory for all patients. All Adverse effects reported during the study period were monitored using a structured questionnaire. The questionnaire consisted of questions about the occurrence of ADR such as diarrhea, nausea and/or vomiting, abdominal pain, metallic taste, symptoms related to an allergic reaction, headache, dizziness or any other undesirable effect.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females (18-65)
2. Diagnosis of primary hypercholesterolemia
3. With total cholesterol 200-239mg/dl and LDL 100-159mg/dl.

Exclusion Criteria:

1. Familial hypoalphalipoproteinemia
2. Patients receiving antihyperlipidemic agents (Statins, Niacin, Fibrates and Bile Sequestrants) were excluded in recent past.
3. Pregnant, breast feeding and women likely to become pregnant
4. Subjects excluded who suffered from allergy or hypersensitivity from Ginger or its tablet excipients.
5. All those subjects excluded with severe or unstable medical conditions like renal failure, Seizures, previous liver surgery, poor controlled diabetes, and drug/alcohol dependence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of total lipid profile | baseline to 2 month
  Change in total cholesterol, triglycerides, High Density Lipoprotein (HDL)Low Density Lipoprotein-cholesterol (LDL) at baseline
  Change from baseline in total cholesterol, triglycerides, High Density Lipoprotein (HDL)Low Density Lipoprotein-cholesterol (LDL) after 2 months
Assessment of cardio protective profile | baseline to 2 month
  Change from baseline in serum glutamic-oxaloacetic transaminase (SGOT), glutamic-pyruvic transaminase (SGPT).

SECONDARY OUTCOMES:
Evaluation of the antioxidant effect | baseline to 2 months
  Change From Baseline in antioxidant markers Superoxide dismutase (SOD), Glutathione peroxidase
Effect on sleep cycle | baseline to 2 months
  To evaluate the sleep patterns by using Insomnia Severity Index (ISI) scale after 2 month
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Effect on C-reactive protein (CRP) | baseline to 2 months
  Change From Baseline in antioxidant marker C-reactive protein (CRP)
Effect on memory | baseline to 2 months
  Change in memory enhancement effect through mini mental state examination (MMSE) scale at baseline and after 2 months
  The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be memory impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Alkhidmat Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No